CLINICAL TRIAL: NCT06845358
Title: A Phase 1 Open-Label Human Vaccination and Challenge Study to Assess the Ability of Intradermal BCG TICE(R) Vaccination to Induce Protective TB Immunity Capable of Inhibiting Replication In Vivo in Healthy Human Volunteers
Brief Title: Safety and Challenge Study of BCG TICE(R) Vaccination to Test Tuberculosis Immunity in Heathy Humans
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study not implemented due to funding.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 22-0011; 5UM1AI148684-03 (NIH)
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05-15

CONDITIONS: Tuberculosis
Keywords: BCG Vaccination; Intradermal; Open-label; Phase 1; Protective Immunity; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — BCG Vaccine; Sodium Chloride; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Subjects will receive 0.1 mL dose of 2x10^6 colony-forming units (CFU) Bacille Calmette-Guerin (BCG) TICE (R) vaccine, administered intradermally over the deltoid muscle of the preferred arm on Day 1. Subjects will then be challenged with 0.1mL of 4x10^6 colony-forming units (CFU) Bacille Calmette-Guerin (BCG) TICE (R) administered intradermally 6 months after vaccination. N=32
  Interventions: Biological: BCG TICE strain; Other: Sodium Chloride, 0.9%; Other: Sterile Water for Injection
- Arm 2 (Experimental): Subjects will receive a 0.1mL dose of 4x10^6 colony-forming units (CFU) Bacille Calmette-Guerin (BCG) TICE (R) administered intradermally over the deltoid muscle of the preferred arm after complete enrollment of Arm 1 subjects. N=32
  Interventions: Biological: BCG TICE strain; Other: Sodium Chloride, 0.9%; Other: Sterile Water for Injection

INTERVENTIONS:
Biological: BCG TICE strain — BCG TICE strain is an attenuated, live culture preparation of the BCG strain of Mycobacterium bovis.
Other: Sodium Chloride, 0.9% — 0.9% Sodium Chloride Injection
Other: Sterile Water for Injection — A sterile, nonpyrogenic preparation of water for injection which contains no bacteriostat, antimicrobial agent or added buffer and is supplied only in single-dose containers to dilute or dissolve drugs for injection

SUMMARY:
A nonrandomized, open-label trial will be conducted with a total of 64 healthy male and non-pregnant females, ages 18-45 years. Participants in Group A will enroll 32 participants to receive 2x10^6 colony- forming units CFU TICE(R) BCG vaccination on Day 1 and 4x10^6 CFU challenge on Day 181. Once enrollment has been completed in Group A, participants in Group B will be enrolled sequentially to receive 4x10^6 CFU challenge. The primary objectives are to evaluate the safety of intradermal (ID) TICE(R) BCG for use as a human challenge model for Mycobacterium tuberculosis (Mtb) infection and to examine BCG shedding from challenge sites in participants who had received ID vaccination with TICE(R) BCG or were not vaccinated six months prior.

DETAILED DESCRIPTION:
A nonrandomized, open-label trial will be conducted with a total of 64 healthy male and non-pregnant females, ages 18-45 years. Participants in Group A will enroll 32 participants to receive 2x10^6 colony- forming units (CFU) TICE(R) BCG vaccination on Day 1 and 4x10^6 CFU challenge on Day 181. Once enrollment has been completed in Group A, participants in Group B will be enrolled sequentially to receive 4x10^6 CFU challenge. The primary objectives are to evaluate the safety of intradermal (ID) TICE(R) BCG for use as a human challenge model for Mycobacterium tuberculosis (Mtb) infection and to examine BCG shedding from challenge sites in participants who had received ID vaccination with TICE(R) BCG or were not vaccinated six months prior. The secondary objectives are to 1) evaluate the safety of ID TICE(R) BCG after vaccination, 2) examine BCG shedding by MGIT assay from challenge sites in participants who had received ID vaccination with TICE(R) BCG or were not vaccinated six months prior, 3) examine BCG shedding from challenge sites in participants that had received ID vaccination with TICE(R) BCG or were not vaccinated six months prior using additional assays, 4) characterize the T cell responses after BCG challenge in participants that received ID vaccination with TICE(R) BCG or not vaccinated six months prior and 5) determine whether IFN-gamma correlates with levels of BCG shedding.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Stated willingness to be available for all study visits and comply with all trial procedures throughout the duration of the trial.
3. Are males or non-pregnant females between the ages of 18 and 45 years, inclusive, at the time of enrollment.
4. For women of childbearing potential, negative serum pregnancy test at screening and negative urine pregnancy test within 24 hours prior to vaccination and challenge of TICE(R) BCG.

   Women of childbearing potential*Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy, or < 1 year of the last menses if menopausal.

   **Must agree to use highly effective contraception (defined as those that result in a failure rate with correct use of less than 1 percent per year) from 30 days prior to receipt of the first dose of investigational product until at least 3 months after receipt of the last administration.

   ***Includes the following methods used alone: bilateral tubal ligation/bilateral salpingectomy, intrauterine system (IUS)/intrauterine device (IUD), estrogen/progestin-only oral, injectable, and implantable contraceptives, and abstinence when it is a consistent lifestyle choice.

   ****The following methods must be used together: male condom with a female non-condom barrier method (including diaphragm, cervical cap, contraceptive sponge, vaginal spermicide), female condom with diaphragm, cervical cap, contraceptive sponge, vasectomy with female barrier method (including female condom, diaphragm, cervical cap, contraceptive sponge, vaginal spermicide).
5. Are in good health, as judged by the investigator and determined by vital signs, medical history, physical examination, and safety labs within normal range*****.

   *****Oral temperature, pulse rate (PR), and blood pressure (BP), medical history, physical examination, and safety labs within normal ranges (except creatinine and alanine transaminase [ALT] levels below the normal ranges that will not be considered clinically significant abnormalities). Baseline screening labs should fall within the normal range of the clinical reference lab.
6. Have a negative HIV-1 ELISA test at first screening visit.
7. Have negative serology tests for hepatitis B surface antigen and hepatitis C virus antibody at first screening visit.
8. Have a negative QuantiFERON(R) - (tuberculosis)TB Gold test at first screening visit..
9. Have a urine dipstick that is negative for glucose and is less than 1 for protein at all screening visits.
10. Ability to understand and complete all study visits as required per protocol and be reachable by telephone.
11. Male participants must refrain from donating sperm from the screening visit until at least 12 weeks after the last administration.

Exclusion Criteria:

1. Have a history of suspected, confirmed, treated, or have other evidence of active tuberculosis, including a positive PPD skin test*

   *Symptoms of pulmonary tuberculosis (TB) may include productive cough for more than two or three weeks in duration, lymphadenopathy, fever, night sweats, unintentional weight loss in a person with known or possible TB exposure, and/or past or present residence in or travel to an area where TB is endemic.
2. Have any systemic symptoms within 72 hours prior to BCG administration or signs of acute febrile illness (AFI) or acute respiratory illness (ARI)**

   **(e.g., fever, cough, rhinorrhea, etc.) before TICE(R) BCG administration or signs of lymphadenopathy, hepatosplenomegaly, or pulmonary disease by physical exam on day of TICE(R) BCG administration.
3. Have history of any significant acute or chronic medical conditions related to immunosuppression***.

   ***Such as impaired immunocompromised state due to chronic or acute disease or receipt of immunosuppressant drugs or therapies, including steroids, alkylating agents, antimetabolites, or radiation.
4. Chronic medications that, in the opinion of the investigator, will interfere with immunity or affect safety.
5. Receipt of >/= 20 milligrams (mg)/day of prednisone or equivalent for >/= 14 consecutive days in a four-week period prior to signing the informed consent.
6. Have any history of excessive scarring or keloid formation.
7. Have household contact or occupation involving significant close contact, such as living with or directly working with someone who is immunocompromised.
8. Have a pacemaker, prosthetic valve, or implantable cardiac devices, endovascular grafts, prosthetic joint implants, intramedullary nails, or titanium brain implants.
9. Have a known allergy to any TICE(R) BCG components.
10. Received blood products or immunoglobulin within six months prior to TICE(R) BCG administration.
11. Received immunotherapy within one year prior to TICE(R) BCG administration.
12. Received or plan to receive live attenuated vaccines four weeks before or after TICE(R) BCG administration.
13. Received or plan to receive inactivated or killed vaccines two weeks before or after TICE(R) BCG administration.
14. Plans to enroll in another clinical trial that could interfere with safety assessment of the study product at any time during the study period.
15. Received an experimental agent within 30 days prior to TICE(R) BCG administration or planned receipt of an experimental agent within 90 days after TICE(R) BCG administration.
16. Have a history of use of a systemic antibiotic within 14 days prior to TICE(R) BCG administration or planned use of a systemic antibiotic within three months after TICE(R) BCG administration.
17. Anyone working as a healthcare provider during the trial.
18. Are breastfeeding or plan to breastfeed at any given time throughout the study.
19. Have a history of alcohol or drug abuse in the last five years.
20. Have a BMI < 18.5 or >/= 35.
21. Current or history of eczema and psoriasis.
22. Received prior BCG vaccination (prior to participation in this study).
23. History of infection with pulmonary or extrapulmonary Nontuberculous Mycobacteria (NTM).
24. Currently living with someone or in close contact with someone with active TB.
25. PPD skin test within two months prior to TICE(R) BCG administration or receipt during the study.
26. Participants who meet eligibility criteria for Group A, but decline will not be eligible to enroll in Group B.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11-26 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of the area under the curve (AUC) for repeated measures of shedding over time from mycobacteria growth indicator tube (MGIT) BACTEC assays after intradermal (ID) TICE (R) Bacille Calmette-Guerin (BCG) challenge | Day 185 through Day 237
Serious adverse events (SAE) and/ or Medically Attended Adverse Events (MAAEs) related to intradermal (ID) TICE (R) Bacille Calmette-Guerin (BCG) challenge | Day 181 through Day 361
The number of participants experiencing Grade 3 (severe) or higher clinical safety laboratory adverse events (AEs) following intradermal (ID) TICE(R) Bacille Calmette-Guerin (BCG) challenge | Day 181 through Day 188
The number of participants experiencing Grade 3 (severe) or higher solicited injection site reactions following intradermal (ID) TICE(R) Bacille Calmette-Guerin (BCG) challenge | Day 181 through Day 236
The number of participants experiencing Grade 3 (severe) or higher solicited systemic reactions following intradermal (ID) TICE(R) Bacille Calmette-Guerin (BCG) challenge | Day 181 through Day 195
The number of participants reporting Grade 3 (severe) or higher adverse events (AEs) related to intradermal (ID) TICE (R) Bacille Calmette-Guerin (BCG) challenge | Day 181 through Day 237

SECONDARY OUTCOMES:
Analyze the adaptive immune responses associated with immunogenicity and reactogenicity | Day 181 through Day 279
  Measured using IFN-gamma ELISPOT assay
Comparison of area under the curve (AUC) for repeated measures of shedding over time from MGIT BACTEC assays intradermal (ID) TICE (R) Bacille Calmette-Guerin (BCG) challenge between unvaccinated and vaccinated groups. | Day 4 through Day 57
Distribution of the area under the curve (AUC) for repeated measures of shedding over time from colony-forming units (CFU) assays after intradermal (ID) TICE (R) Bacille Calmette-Guerin (BCG) challenge. | Days 4 through Day 57
Distribution of the area under the curve (AUC) for repeated measures of shedding over time from quantitative reverse transcription polymerase chain reaction (qRT-PCR) assays after intradermal (ID) TICE (R) Bacille Calmette-Guerin (BCG) challenge. | Days 4 through Day 57
Medically Attended Adverse Events (MAAEs) and Serious adverse events related to intradermal (ID) TICE (R) Bacille Calmette-Guerin (BCG) administration after vaccination | Day 1 through Day 181
Test correlations between interferon gamma (IFN-gamma) ELISPOT responses and Bacille Calmette-Guerin (BCG) shedding | Day 181 through Day 279
The number of participants experiencing Grade 3 (severe) injection site reactions following intradermal (ID) TICE (R) Bacille Calmette-Guerin (BCG) vaccination. | Day 1 through Day 30
The number of participants experiencing Grade 3 (severe) or higher clinical safety laboratory adverse events (AEs) following intradermal (ID) TICE (R) Bacille Calmette-Guerin (BCG) vaccination. | Day 1 through Day 181
The number of participants experiencing Grade 3 (severe) or higher solicited systemic reactions following intradermal (ID) TICE (R) Bacille Calmette-Guerin (BCG) vaccination. | Day 1 through Day 30
The number of participants reporting Grade 3 (severe) or higher adverse events (AEs) related to intradermal (ID) TICE (R) Bacille Calmette-Guerin (BCG) vaccination | Day 1 through Day 57